CLINICAL TRIAL: NCT07102212
Title: Randomized Clinical Trial of a Telemedicine-mHealth Symptom Cluster Intervention for Advanced Cancer Patients: Increasing Access in Rural Areas
Brief Title: Telemedicine-mHealth Symptom Cluster Intervention for Advanced Cancer Patients: Finding Our Center Under Stress (FOCUS)
Acronym: FOCUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Ohio University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharla Wells-Di Gregorio, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OSU-24212; NCI-2025-05185 (Other: CTRP (Clinical Trial Reporting Program)); R01CA281885 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-08-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Breast Cancer; Prostate Cancer; Multiple Myeloma; Melanoma
Keywords: symptom management; cancer; rural; sleep; anxiety; worry; fatigue; mood; depression; mHealth; telemedicine; app; advanced cancer; Appalachian
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Multiple Myeloma; Melanoma; Neoplasms; Anxiety Disorders; Fatigue; Depression; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The overall goal of this randomized clinical trial is to evaluate the effectiveness of a telemedicine-mHealth symptom cluster intervention, Finding Our Center Under Stress (FOCUS), with people with advanced cancer. The investigators include a telemedicine-mHealth information control condition for comparison.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a prospective, tripleblind (i.e., patient, research assistant, statistician), single-site, randomized, clinical effectiveness trial of a brief, tailored, minimal contact telemedicine-mHealth symptom management intervention for people with advanced cancer from rural areas.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOCUS Intervention Arm (Experimental): FOCUS is a standardized mHealth-integrated CBT-ACT biobehavioral intervention divided into four modules. FOCUS includes an introductory video, sleep diary, app overview and a sleep module, worry-uncertainty module, fatigue module, and a mood module (each 1.5 hours spread over a week), for a total of 6 hrs of direct mHealth intervention (not including home practice time) spaced across 6 wks. All modules include behavioral and values-based exercises. The app also features motivational features/rewards for skill-based home practice activities. FOCUS Telemedicine Component. Psychosocial Oncology Fellows (Ph.D. clinical psychologists) will provide minimal contact professional support, connecting with participants via telemedicine for 15-20 min each week to answer questions about skills and home practice after each module. Our project coordinator will respond to any technical or study issues with Moby support, our mobile app design team.
  Interventions: Behavioral: mHealth Intervention
- Information Control Arm (Sham Comparator): Participants will be randomly assigned to an area of the mHealth app specific for control participants. This section of the app will contain a similar video introduction and instructions for use of the app followed by four symptom modules - sleep, worry, fatigue, and mood containing standardized patient information from NCI for each symptom. Control Group Telemedicine Component. Participants will receive weekly minimal contact with a postdoctoral fellow who will assess understanding of NCI symptom management materials with standardized questions focused on that week's material, note information to be reviewed the following week, answer any study-related questions, and record any symptom management practices initiated since reviewing these materials.
  Interventions: Behavioral: mHealth Intervention

INTERVENTIONS:
Behavioral: mHealth Intervention — Participants are randomized to the FOCUS app or Information Control section of the app and will have six weeks to complete the app. Randomization, via the app, is stratified by geographic location (rural vs other), cancer type, and demographics so experimental arms are equivalent. Participants will complete 5 assessments online over a 12-mo period. The participants will have weekly telehealth professional support during the six-week intervention. Participants wear GeneActiv watches for sleep/activity recording for 7 days and provide blood and saliva samples at baseline, 6 and 12 weeks, and 6 and 12 months.

SUMMARY:
In response to the symptom needs experienced in advanced cancer, the investigators developed a brief, integrated CBT-ACT symptom management intervention, Finding Our Center Under Stress (FOCUS). Using FOCUS, participants learn skills to self-manage sleep, worry-anxiety, depression, and fatigue and improve their ability to focus on what matters most to them despite these symptoms. Results of the pilot randomized controlled trial with people with advanced cancer demonstrate improved sleep on both self-report and physiologic (i.e., actigraphy) measures, and improvements on worry, depression, and fatigue interference with strong effect sizes ranging from d= 0.59 to 0.98 and sleep effects 12 months post-treatment. The investigators refined the fatigue module with exercise modifications and beta-tested the FOCUS intervention as an mHealth web-based app for acceptability with 10 diverse patients with advanced cancer -100% would recommend for other advanced cancer patients. The overall objective of this proposed randomized effectiveness trial is to evaluate the impact of this telemedicine-mHealth symptom cluster intervention with patients from rural and Appalachian communities (where the PI was raised). Innovative features include a focus on a symptom cluster including anxiety, integrated CBT-ACT intervention, telemedicine-mHealth delivery method, and biobehavioral approach evaluating behavioral and inflammatory mediators.

DETAILED DESCRIPTION:
The investigators will deliver an evidence-based intervention for a common cancer symptom cluster, with clinically significant pilot findings, to rural, underserved people with advanced cancer. The investigators will improve access via a telemedicine- mHealth approach, developed and refined based on the needs and evaluative feedback of people with advanced cancer. The investigators aim to reduce symptom severity and interference via an integrated CBT-ACT intervention. In addition, the investigators will examine the behavioral, hormonal, and inflammatory mechanisms of symptom change including several novel biomarkers identified in the pilot trial (e.g., IL-12, IL-1alpha, TNFbeta). An effective, accessible, brief alternative to medication-based symptom cluster management is essential given the limited availability of palliative and psychosocial care for this population and impact of these symptoms on patient functional status, quality of life, treatment adherence, and survival. The study aligns with NCI's goal to enhance access to clinical trials via telemedicine and mobile applications to better meet the survivorship needs of underserved populations and the goal of RFA CA-22-027 to test interventions to improve delivery of comprehensive survivorship care for individuals with advanced cancer.

SPECIFIC AIMS:

Aim 1: Evaluate the effectiveness of a telemedicine-mHealth symptom management intervention (FOCUS) targeting a common symptom cluster for people with advanced cancer

Aim 2: Determine the impact of FOCUS dose on symptom severity and interference and examine usage by patient geographic location and other demographics

Aim 3 (Exploratory): Examine biobehavioral mediators of treatment effects

ELIGIBILITY:
Inclusion Criteria:

* Participants will include 120 people with advanced cancer who are ≥ 18 yrs old
* Able to read and write in English
* Who use internet and e-mail as determined by Computer & Mobile Device Proficiency Questionnaire.
* People with stage IIIb&c/IV lung cancer, stage IV breast cancer, stage IV prostate cancer, advanced (on active treatment) multiple myeloma, and stage IIIb & IV melanoma (24 of each cancer type)
* meet clinical cut-offs on any two symptoms in this cluster (i.e., ≥ 8 on Insomnia Severity Index (ISI), ≥ 3 on Patient Health Questionnaire-2 for depression, ≥ 2 on Generalized Anxiety Disorder-2, ≥ 3 on Fatigue Symptom Inventory Severity)

Exclusion Criteria:

* Night-shift work
* Untreated bipolar disorder
* Substance use disorder
* Cognitive impairment per Brief Screen for Cognitive Impairment
* Eastern Cooperative Oncology Group performance status of 3 or greater (in bed 50% or more of day), or <6 mos predicted survival per oncology team.
* Prior participation in cognitive behavior therapy will not be an exclusion criterion if individuals meet symptom severity threshold for at least two symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline, 6 and 12 weeks, and 6 and 12 months
  Symptom measures of insomnia will be made using the Insomnia Severity Index, a scale from 0 to 28 with higher scores indicating greater insomnia
Center for Epidemiological Studies Depression Scale | Baseline, 6 and 12 weeks, and 6 and 12 months
  Symptom measures of depression will be made using the Center for Epidemiological Studies Depression Scale, a scale from 0 to 60 with higher scores indicating more depressive symptoms/more severe depression
Fatigue Severity Index | Baseline, 6 and 12 weeks, and 6 and 12 months
  Symptom measures of fatigue will be made using the Fatigue Severity Index, a scale from 0 to 110 with higher scores indicating more severe fatigue
Generalized Anxiety Disorder | Baseline, 6 and 12 weeks, and 6 and 12 months
  Symptom measures of generalized anxiety will be made using the Generalized Anxiety Disorder - 7 (GAD-7), a scale from 0 to 21with higher scores indicating more severe anxiety
App Dose and Use | Up to 12 months
  The investigators will analyze usage reports of participant engagement with FOCUS mHealth application to assess time reviewing the four FOCUS modules (sleep, worry, depression, fatigue) and overall time using the application to evaluate dose-response on symptoms. The investigators will compare FOCUS usage by geographic location (rural vs other) and demographics and complete detailed examination of clickmaps, screen recordings, and module usage.
Symptom Interference/Quality of Life | Baseline, 6 and 12 weeks, 6 and 12 months
  The investigators will use the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) five functional sub-scales to assess symptom interference. The subscales will be totaled and the overall scale will range from 0 to 110 with higher scores on functional scales and global health status/quality of life representing better functioning.

SECONDARY OUTCOMES:
Biobehavioral Mediators | Baseline, 6 and 12 weeks, and 6 and 12 months
  The investigators will test whether symptom severity is mediated by stress hormones (cortisol) and inflammation (IL-12, IL-1alpha, IL-1beta, TNF-alpha, TNFbeta, IL-6, hsCRP, exotaxin) by measuring the levels of each biomarker at various time points throughout the study.
CAQ-8 (Committed Action Questionnaire) | Up to 12 months
  The investigators will test whether symptom severity is mediated by behavioral changes (committed action - Committed Action Questionnaire). The CAQ-8 scale ranges from 0 to 48 with higher levels indicating a more committed action.
AAQ-II (Acceptance and Action Questionnaire) | Up to 12 months
  The investigators will test whether symptom severity is mediated by behavioral changes (psychological flexibility - Acceptance and Action Questionnaire). The AAQ-II scale ranges from 7 to 49 with higher scores representing greater psychological inflexibility. This measure will be reverse scored so that higher scores represent greater psychological flexibility to test the mediator hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Sharla Wells-Di Gregorio, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NIH Data Sharing Policy, data from this project, including questionnaire data, de-identified demographics and disease information, as well as biomarker data will be shared at the completion of the study via computerized dataset. The investigators do not plan to release data pertaining to participants' individual web-usage as this data is believed to be private and not essential to the overarching purposes or goals of the project. However, the investigators will release summary statistics pertaining to usage (total app usage, frequency of home practice) so Aim 2 of this study can be evaluated by others interested in the web-usage and descriptive features of the study.
  A study codebook will be provided outlining the methodology and procedures used to collect the data, variable definitions and labels, scored variable information, and information on the general structure/timepoint labeling of the available data.
Supporting Information: SAP, ICF
Time Frame: The investigators will release data in "waves" relating to publications deriving from this data. For instance, our trial sleep data will be released after Aim 1 is published, our immunology data after Aim 3 is published, and all other data will be available after study is completed via Cancer Data Services. Data will remain available for 15 years. After this time, treatment advances may affect how these diseases are treated and/or symptoms are addressed.
Access Criteria: Researchers with certified training in human subjects protections will be able to request access. The investigators will utilize a data sharing agreement that requires 1) a commitment to using the data and codebook only for research purposes, 2) a commitment to securing the data via appropriate computer technology, and 3) a commitment to destroying or returning the data after analyses are complete.
URL: https://psychosocialoncology.wixsite.com/focus

REFERENCES:
- [Background] Wells-Di Gregorio SM, Marks DR, DeCola J, Peng J, Probst D, Zaleta A, Benson D, Cohn DE, Lustberg M, Carson WE, Magalang U. Pilot randomized controlled trial of a symptom cluster intervention in advanced cancer. Psychooncology. 2019 Jan;28(1):76-84. doi: 10.1002/pon.4912. Epub 2018 Oct 30. PMID 30335211
- See also: FOCUS study website — https://psychosocialoncology.wixsite.com/focus
- See also: Information about the James Cancer Hospital and Solove Research Institute — http://cancer.osu.edu